CLINICAL TRIAL: NCT04045275
Title: Feasibility and Preliminary Effects of a Mobile App on Sleep Disturbance
Brief Title: Feasibility of a Mobile App on Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Calm.com, Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer Huberty, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010050
Record Dates: First submitted 2019-07-15; First posted 2019-08-05 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Calmodulin

STUDY DESIGN:
Intervention Model Description: The study design was a randomized control trial with baseline and post-intervention assessments (8 wks from baseline). Individuals reporting sleep difficulties were randomized to either a meditation mobile app intervention (Calm) group or a delayed response group. Participants were randomized after the completion of baseline and informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calm (Experimental): The intervention will occur across 8 weeks. During Week 1, it is suggested to intervention participants that they complete "7 days of Calm" meditation series (7 meditations, each approximately 10 minutes long, created to help users learn the basics of mindfulness meditations. For the remaining weeks (Week 2- Week 8) intervention participants will be asked to meditate for 10 minutes per day using any of the meditation sessions/features. Throughout the intervention, participants not completing 30 minutes of meditation per week will be sent reminders texts/emails.
  Interventions: Behavioral: Calm
- Control (No Intervention): This group is a wait-list control group who will receive the intervention following the 8-week waiting period. Participants in this condition are instructed not to start meditating before the waiting period. After the 8-week waiting period, waitlist participants will receive the same intervention as described in the Calm Arm.

INTERVENTIONS:
Behavioral: Calm — Calm provides daily, 10-minute, guided meditations grounded in mindfulness-based stress reduction (MBSR) and Vipassana meditation. Calm also offers "Sleep Stories," developed using techniques from Cognitive Behavioral Therapy and Relaxation Technique. Clam also includes behavioral components to reinforce sustained practice.
  Arms: Calm

SUMMARY:
This study investigates the feasibility and effects of a mindfulness meditation mobile application on sleep for individuals reporting sleep disturbances.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of a mindfulness meditation mobile application on sleep in individuals reporting sleep disturbances.

The investigator's guiding hypothesis is that the combined elements of a consumer-based mobile meditation app, Calm (e.g., daily mindfulness meditation, sleep stories and behavioral components), will be feasible, accepted and associated with sustained improvement in sleep among individuals who self-identify as having sleep disturbances. Calm provides daily, 10-minute, guided meditations grounded in mindfulness-based stress reduction (MBSR) and Vipassana meditation. Uniquely, Calm also offers "Sleep Stories", developed using techniques from Cognitive Behavioral Therapy and Relaxation Technique.

This is a randomized control feasibility study with an intervention and waitlist control.

Aim 1: Examine the feasibility of using a consumer-based mindful meditation app for >10 mins/day over eight weeks for 100 adults who self-identify as sleep disturbed.

Aim 2: Explore the preliminary effects of Calm on sleep disturbance and emotional symptoms associated with sleep disturbance (i.e. stress, anxiety, depressive symptoms) as compared to those in a wait-list control group.

Recruitment: Participants will be recruited nationally via Internet-based strategies including social media (e.g. Facebook, Twitter, Instagram), social networking sites and email listservs. Recruitment flyers will be posted on social media websites. ResearchMatch.org will be also be utilized as a recruitment tool for this protocol.

Eligibility: Inclusion criteria are: (1) self-identify as sleep disturbed (i.e., score >10 on the Insomnia Severity Index), (2) >18 years of age, (3) English speaking, (4) willing to download the Calm app to their smartphone, and (5) have not practiced meditation more than 60 minutes a month in the past six months (6) willing to be randomized. Participants will report use of medication for sleep at baseline, mid-intervention and post-intervention and not excluded for medication.

Enrollment: Interested participants will complete a brief (5-10 minute) eligibility screener via Qualtrics. Participants will not be made know of sponsor name before randomization assignment to avoid disclosing the app that they will be using. Eligible participants will be asked to sign an electronic informed consent prior to the start of the intervention. After informed consents have been completed, participants (N=100) will be identified. Once eligible participants have been identified, they will be emailed instructions. Ineligible participants will be notified by email.

Tracking: Intervention participants (n=50) usage will be continuously tracked throughout the intervention by Calm.

Post-intervention: Post-intervention questionnaire will be emailed to intervention and control participants via a link from Qualtrics. All participants will have access to Calm after the 8-week study period, but will not be asked to meditate.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as sleep disturbed (i.e., score >10 on the Insomnia Severity Index)
* at least 18 years of age
* English speaking
* willing to download Clam app on their smartphone
* willing to be randomized

Exclusion Criteria:

* have participated in more than 60 minutes of meditation/month within the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Acceptability, as measured by participants' satisfaction with the content in the mindful meditation app | Participant satisfaction is measured immediately after the the conclusion of the 8-week intervention.
  Participants' satisfaction will be measured by participant responses to the item, "On a scale of 1-5 (1=did not enjoy at all, 5=very much enjoyed), how would you rate your overall enjoyment with using Calm (i.e., likeable, pleasurable)?" on an investigator-developed survey. Participants rate their satisfaction on a five-point scale, ranging from 1 (did not enjoy at all) to 5 (very much enjoyed).
Acceptability, as measured by participants' perceptions of the appropriateness of the content in the mindful meditation app | Participants' perceptions of appropriateness are measured immediately after the the conclusion of the 8-week intervention.
  Participants' perceptions of appropriateness will be measured using six items on investigator-developed survey. Items inquire about participants' perceptions regarding the app's ease of use, aesthetics and graphics, and adequacy of the instruction (all rated on 1-5 scales, with higher ratings reflecting greater perceived appropriateness), and three items about the appropriateness of the duration of daily meditations, sleep meditations, and Sleep Stories (rated on a 1-4 scale, with higher ratings reflecting greater perceived appropriateness). Average scores will be reported for each item.
Demand, as assessed by the percentage of participants who use the mindful meditation app for the 70% of the prescribed weekly minutes (≥ 70 minutes/week) | Duration use app use is recorded continuously throughout the 8-week intervention.
  The amount of time that participants use the app will be recorded by Calm (internally) and shared with Arizona State University.
Demand, as assessed by the the comparative frequency of participants use of meditation, sleep meditation, and Sleep Stories | Frequency of use app use is recorded continuously throughout the 8-week intervention.
  The frequency of using individual app components will be recorded by Calm (internally) and shared with Arizona State University.
Demand, as assessed by the the comparative duration of participants use of meditation, sleep meditation, and Sleep Stories | Duration use app use is recorded continuously throughout the 8-week intervention.
  The amount of time that participants use the app individual app components will be recorded by Calm (internally) and shared with Arizona State University.
Preliminary effects of the mindfulness meditation app on sleep disturbance, as assessed by changes in participants' nightly sleep duration over the course of the 8-week intervention period | Sleep diaries are completed daily throughout the 8-week intervention. Each morning, participants report on the previous night's sleep. Participants submit their daily diary entries at the end of each week.
  Sleep duration will be calculated using participants' reports of the time they fell asleep at night, the time that they woke up in the morning, and the amount time spent awake after waking up during the night. These times are self-reported in a gold-standard daily sleep diary.
Preliminary effects of the mindfulness meditation app on sleep disturbance, as assessed by changes in the amount of time required for participants' to fall asleep over the course of the 8-week intervention period | Sleep diaries are completed daily throughout the 8-week intervention. Each morning, participants report on the previous night's sleep. Participants submit their daily diary entries at the end of each week.
  The amount of time required to fall asleep will be measured by participants' self-reports in their daily sleep diaries.
Preliminary effects of the mindfulness meditation app on sleep disturbance, as assessed by changes in the frequency of participants' nightly mid-sleep awakenings over the course of the 8-week intervention period | Sleep diaries are completed daily throughout the 8-week intervention. Each morning, participants report on the previous night's sleep. Participants submit their daily diary entries at the end of each week.
  The frequency of mid-sleep awakenings will be measured by participants' self-reports in their daily sleep diaries.
Preliminary effects of the mindfulness meditation app on sleep disturbance, as assessed by changes in the amount of time spent awake after mid-sleep awakenings over the course of the 8-week intervention period | Sleep diaries are completed daily throughout the 8-week intervention. Each morning, participants report on the previous night's sleep. Participants submit their daily diary entries at the end of each week.
  The amount of time spent awake after mid-sleep awakenings will be measured by participants' self-reports in their daily sleep diaries.
Preliminary effects of the mindfulness meditation app on sleep disturbance, as assessed by changes in participants rating of sleep quality over the course of the 8-week intervention period | Sleep diaries are completed daily throughout the 8-week intervention. Each morning, participants report on the previous night's sleep. Participants submit their daily diary entries at the end of each week.
  Sleep quality will be measured by participants' responses to the question, "How would you rate the quality of your sleep? (1= very poor and 5= very good)," which is included in participants' daily sleep diaries.
Preliminary effects of the mindfulness meditation app on sleep disturbance, as assessed by changes in participants' pre- and post-intervention scores on the Cognitive and Somatic Arousal subscales of the Pre-Sleep Arousal Scale | The Pre-Sleep Arousal Scale will be completed at immediately before (i.e., baseline) and immediately after the intervention
  The Pre-Sleep Arousal Scale is a 16-item self-report questionnaire that measures arousal before sleep. Items describe symptoms of cognitive and somatic arousal. Using a five-point scale (1, not at all; 2, slightly: 3, moderately; 4, a lot; 5, extremely), participants rate extent to which they generally experience each symptom as they attempt to fall asleep. The Pre-Sleep Arousal Scale is comprised of two eight-item subscales, which assess Cognitive Somatic arousal. Subscale scores are determined by summing ratings from the included items. Possible scores on each subscale range from 8 to 40, with higher scores indicating greater pre-sleep arousal.
Preliminary effects of the mindfulness meditation app on sleep fatigue, as assessed by changes in participants' pre- and post-intervention scores on the Fatigue Severity Scale | The Fatigue Severity Scale will be completed at immediately before (i.e., baseline) and immediately after the intervention
  The Fatigue Severity Scale is a nine-item self-report measure of fatigue and the extent to which fatigue interferes with daily living. Respondents rate the extent to which they agree with statements about their experience with fatigue during the past week. Items are scored on a seven-point scale ranging from 1 to 7 (1=strongly disagree, 7=strongly agree). Total scores range from 1 to 7, reflecting the mean rating of the items. Higher scores indicate greater fatigue.
Preliminary effects of the mindfulness meditation app on sleepiness, as assessed by changes in participants' pre- and post-intervention scores on the Epworth Sleepiness Scale | The Epworth Sleepiness Scale will be completed at immediately before (i.e., baseline) and immediately after the intervention
  The Epworth Sleepiness Scale is an eight-item measure of daytime sleepiness. Respondents use a four-point scale to rate the likeliness that they would doze off or fall asleep in eight situations involving activities with low levels of stimulation, relative immobility, and relaxation, based on their usual way of life in recent times. Item ratings range from 0 to 3 (0=would never doze, 3=high chance of dozing). Items are summed to calculate a total score, ranging from 0 to 24, with higher scores indicating greater sleepiness.

SECONDARY OUTCOMES:
Preliminary effects of the mindfulness meditation app on depression, as assessed by changes in participants' pre- and post-intervention scores on the Depression Anxiety Stress Scale-21 Items | The Depression Anxiety Stress Scale-21 Items will be completed at immediately before (i.e., baseline) and immediately after the intervention
  The Depression Anxiety Stress Scale-21 Items is a set of three seven-item self-report scales measuring depression, anxiety, and stress/tension. Respondents use a four-point scale, ranging from 0 to 3, to rate the extent to which symptoms of depression, anxiety, and stress apply to their experiences during the past week (0=did not apply to me at all, 3=applied to me very much, or most of the time). For each scale, ratings for the relevant items are summed, and sums for each scale are multiplied by two to allow for comparison with scores from the original the 42-item version of the Depression Anxiety Stress Scale; thus total scores range from 0 to 42, with higher scores indicating greater depression, anxiety, and stress.
Preliminary effects of the mindfulness meditation app on depression, as assessed by changes in participants' pre- and post-intervention scores on the Hospital Anxiety and Depression Scale | The Hospital Anxiety and Depression Scale will be completed at immediately before (i.e., baseline) and immediately after the intervention
  The Hospital Anxiety and Depression Scale is a 14-item questionnaire, comprised of two seven-item subscales measuring depression and anxiety. Respondents rate the frequency or severity of anxious and depressive symptoms on a four-point scale. Item ratings range from 0 to 3, with higher ratings reflecting more frequent or severe symptoms. Items from each subscale are summed to calculate total scores for depression and anxiety.
Preliminary effects of the mindfulness meditation app on anxiety, as assessed by changes in participants' pre- and post-intervention scores on the Depression Anxiety Stress Scale-21 Items | The Depression Anxiety Stress Scale-21 Items will be completed at immediately before (i.e., baseline) and immediately after the intervention
  The Depression Anxiety Stress Scale-21 Items is a set of three seven-item self-report scales measuring depression, anxiety, and stress/tension. Respondents use a four-point scale, ranging from 0 to 3, to rate the extent to which symptoms of depression, anxiety, and stress apply to their experiences during the past week (0=did not apply to me at all, 3=applied to me very much, or most of the time). For each scale, ratings for the relevant items are summed, and sums for each scale are multiplied by two to allow for comparison with scores from the original the 42-item version of the Depression Anxiety Stress Scale; thus total scores range from 0 to 42, with higher scores indicating greater depression, anxiety, and stress.
Preliminary effects of the mindfulness meditation app on anxiety, as assessed by changes in participants' pre- and post-intervention scores on the Hospital Anxiety and Depression Scale | The Hospital Anxiety and Depression Scale will be completed at immediately before (i.e., baseline) and immediately after the intervention
  The Hospital Anxiety and Depression Scale is a 14-item questionnaire, comprised of two seven-item subscales measuring depression and anxiety. Respondents rate the frequency or severity of anxious and depressive symptoms on a four-point scale. Item ratings range from 0 to 3, with higher ratings reflecting more frequent or severe symptoms. Items from each subscale are summed to calculate total scores for depression and anxiety.
Preliminary effects of the mindfulness meditation app on stress, as assessed by changes in participants' pre- and post-intervention scores on the Depression Anxiety Stress Scale-21 Items | The Depression Anxiety Stress Scale-21 Items will be completed at immediately before (i.e., baseline) and immediately after the intervention
  The Depression Anxiety Stress Scale-21 Items is a set of three seven-item self-report scales measuring depression, anxiety, and stress/tension. Respondents use a four-point scale, ranging from 0 to 3, to rate the extent to which symptoms of depression, anxiety, and stress apply to their experiences during the past week (0=did not apply to me at all, 3=applied to me very much, or most of the time). For each scale, ratings for the relevant items are summed, and sums for each scale are multiplied by two to allow for comparison with scores from the original the 42-item version of the Depression Anxiety Stress Scale; thus total scores range from 0 to 42, with higher scores indicating greater depression, anxiety, and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huberty JL, Green J, Puzia ME, Larkey L, Laird B, Vranceanu AM, Vlisides-Henry R, Irwin MR. Testing a mindfulness meditation mobile app for the treatment of sleep-related symptoms in adults with sleep disturbance: A randomized controlled trial. PLoS One. 2021 Jan 7;16(1):e0244717. doi: 10.1371/journal.pone.0244717. eCollection 2021. PMID 33411779